CLINICAL TRIAL: NCT03348475
Title: Binge Focused Therapy: Examining an Accessible, Cost-effective, Guided, Self-help, Group-based Approach for the Treatment of Binge Eating Disorder
Brief Title: Binge Focused Therapy: A Guided, Self-help, Group-based Approach for Binge Eating Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nova Scotia Health Authority (Other)
Responsible Party: Principal Investigator, Aaron Keshen, Psychiatrist, Nova Scotia Health Authority
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BFT
Record Dates: First submitted 2017-11-16; First posted 2017-11-21 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Binge-Eating Disorder; Eating Disorder
Keywords: Guided self-help; Group-based intervention; Binge Focused Therapy; Brain Over Binge; Non-expert guided; Minimally intensive
MeSH Terms: conditions — Binge-Eating Disorder; Feeding and Eating Disorders | interventions — Methods

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental Group (Experimental): Binge Focused Therapy (BFT) Intervention
  Interventions: Behavioral: Binge Focused Therapy (BFT) Intervention

INTERVENTIONS:
Behavioral: Binge Focused Therapy (BFT) Intervention — The intervention, Binge Focused Therapy, is a 3-session, 8-week, non-expert guided self-help program. Participants will attend sessions at Week 1, Week 2, and Week 8 at the Nova Scotia Health Authority Eating Disorder Clinic. Each session will be approximately 2 hours in length.

SUMMARY:
The "Brain Over Binge Recovery Guide" (Hansen, 2016), is a self-help approach that incorporates fundamental aspects of Acceptance and Commitment Therapy, Dialectical Behavioural Therapy, Motivational Enhancement Therapy and addictions treatment. This approach has been streamlined into a guided self-help protocol (Binge Focused Therapy, or BFT) that can be delivered by undergraduate students with minimal mental health experience in 3 group sessions spread over 8 weeks (i.e., Week 1, Week 2, Week 8). The aim of this proof-of-concept study is to provide preliminary data to examine whether this approach is feasible and has clinical potential for patients with binge eating disorder.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older;
* Meets DSM-5 criteria for moderate to severe Binge Eating Disorder (BED) as determined through screening interview by an eating disorder psychiatrist and validated with the Eating Disorder Diagnostic Scale (a self-report screening tool);
* Provides written informed consent.

Exclusion Criteria:

* Currently receiving treatment for BED;
* Is taking a psychotropic medication (e.g., antidepressant, stimulant, etc.) AND the dose has been changed 2 weeks prior to baseline;
* Insufficient knowledge of English.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2019-10-03 (Actual); Study Completion 2019-10-03 (Actual)

PRIMARY OUTCOMES:
Change in Binge Eating Frequency | Baseline, Week 8, 1-year follow-up
  Self-reported binge eating frequency will be assessed with the Eating Disorder Examination Questionnaire 6.0 (EDE-Q). Binge eating frequency is measured on item 15 of the EDE-Q.

SECONDARY OUTCOMES:
Change in Binge Eating Severity | Baseline, Week 2, Week 8, 1-year follow-up
  Self-reported binge eating severity will be assessed with the Binge Eating Scale (BES). The BES is a 16-item measure, each item has 3-4 coded responses. The total score ranges from 0-46, where a higher score indicates greater binge eating severity.
Remission Rate | Week 8, 1-year follow up
  Remission defined as 100% reduction in binge episodes in the last 28 days of treatment phase preceding week 8, or in the last 28-days of follow-up phase.
Response Rate | Week 8, 1-year follow up
  Responders defined as ≥ 50% reduction in the number of binge episodes from baseline to either of the last two preceding weeks of treatment or follow-up.
Change in General Eating Disorder Symptomatology | Baseline, Week 8, 1-year follow-up
  Self-reported general eating disorder symptomatology will be assessed using the global score generated from the EDE-Q. The EDE-Q is a 28-item measure that assesses four areas of eating disorder psychopathology (eating concern, shape concern, weight concern, dietary restraint). Each item uses a Likert scale ranging from 0 (lowest frequency/severity) to 6 (highest frequency/severity). The global score ranges from 0-6 where higher scores indicate greater impairment. The global score is obtained using the mean of the four subscales.
Change in Locus of Control of Behaviour | Baseline, Week 2, Week 8, 1-year follow-up
  Self-reported locus of control of behaviour will be assessed using the Locus of Control of Behaviour scale (LCB). The LCB scale is a 17-item measure. Participants respond to each item using a Likert scale ranging from 0 (strongly disagree) to 5 (strongly agree). Total scores range from 0-85, with higher scores indicating a greater degree of externality.
Change in Coping Self-Efficacy | Baseline, Week 2, Week 8, 1-year follow-up
  Self-reported coping self-efficacy will be assessed using the Coping Self-Efficacy Scale (CSES). The CSES is a 26-item measure. Each item with be rated using a Likert scale from 1 (cannot do at all) to 10 (certain can do). An average score will be obtained. Higher scores indicate greater coping self-efficacy.
Motivation/Confidence/Readiness for Behaviour Change | Baseline and Week 2
  This will be measured using responses to three Likert-style questions that assess the perceived value of changing binge eating, confidence in ability to change binge eating, and readiness to change binge eating. Each item will be scored on a scale of 1 (not at all important/confident/ready) to 10 (extremely important/confident/ready). Each item will be assessed independently. Higher scores indicate greater motivation, confidence, and readiness.
Depression, Anxiety and Tension/Stress | Baseline
  Self-reported depression, anxiety, and tension/stress will be assessed using the Depression Anxiety Stress Scale (DASS). Participants will respond to 21-items each scored on a Likert scale from 0 (did not apply) to 3 (applied very much or most of the time). A total score ranges from 0-126 with a higher score indicating greater impairment.
Participant Satisfaction with Intervention | Week 8
  Participants will respond to 3 Likert-style questions on a scale of 1 (very poor) to 6 (excellent) and several open-ended questions asking about their perceptions of the program. Higher scores indicate greater satisfaction.
Week 3 - 7 Adherence | Week 8
  Participants' adherence to tracking binge frequency and use of defusion skills (i.e., Homework) between Sessions 2 and 3.

CONTACTS AND LOCATIONS:
Locations (1):
- Nova Scotia Health Authority, Halifax, Nova Scotia, Canada